CLINICAL TRIAL: NCT03975127
Title: Cervical Cytology - Do SMS Reminders Increase Participation in the Cervical Screening Programme?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: GN201905PH
Record Dates: First submitted 2019-05-22; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-05

CONDITIONS: Cervical Carcinoma; Cervical Dysplasia
Keywords: population screening
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Intervention Model Description: The study arms are as follow:
  1. No intervention: women will routinely be invited to attend for cervical screening via the SCCRS application.
  2. Experimental: Women aged under 30 years will be identified to receive an SMS following cervical screening invitation using information from the CHI Broadcast
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine (No Intervention): women will routinely be invited to attend for cervical screening via the SCCRS application.
- SMS (Experimental): Women aged under 30 years will be identified to receive an SMS following cervical screening invitation using information from the CHI Broadcast
  Interventions: Other: SMS text

INTERVENTIONS:
Other: SMS text — A single SMS text sent to women under 30 who are eligible for the cervical screening programme and who have been invited by letter
  Arms: SMS

SUMMARY:
This study will pilot production and evaluate the use of reminder information in women invited for cervical screening for the first time within the GGC eligible population for cervical screening. Women aged under 30 years will be identified to receive an SMS text message following their cervical screening invitation using information from the CHI Broadcast.

DETAILED DESCRIPTION:
Cervical cancer is the commonest cancer among women aged less than 35 years. A change to the age range and frequency for cervical screening was implemented on the 6th June 2016. This increased the younger eligible age for screening from 20 to 25. Uptake of cervical screening among women in the youngest eligible age range has historically been low. Research by Scott Porter has shown that cervical screening is not on young women's radar and additionally there is scope for confusion amongst women in this cohort about the requirement to attend for cervical screening if they have been previously immunised against HPV (human papilloma virus) generally in secondary school in year 2, some 12 years earlier.

The HPV vaccine was introduced in 2008 and is designed to protect against the two types of high risk HPV which cause approximately 75% of all cervical cancer. Advice to all eligible women who have been vaccinated remains that participation in cervical screening is necessary to provide the most comprehensive protection against cervical cancer, as the current vaccine does not provide protection against all high risk cancer causing strains of HPV.

Research from other screening programmes has also shown that where individuals engage with a screening programme from the start, they are more likely to continue to participate in screening for as long as they are eligible.

"Intending to, but not getting round to it", is the reason most associated with non-response to cervical cancer screening invitations.

GGC serves approximately 40% of the total Scottish population and therefore testing the reminder in the GGC population provides an opportunity to compare the impact of the SMS text reminder in this cohort with management as usual within the remainder of the Scottish eligible population. This should enable us to identify whether use of a reminder SMS text message is in fact likely to add value and increase participation in cervical screening.

ELIGIBILITY:
Inclusion Criteria:

* All women aged under 30 years who are eligible for cervical screening with a CHI number and registered with a GP in the NHS Greater Glasgow and Clyde area.

Exclusion Criteria:

* Women have do not have a cervix

Ages: 22 Years to 29 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50000 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Attendance | 12 months
  Number of women attending for cervical screening in intervention group compared to control group

SECONDARY OUTCOMES:
Scottish Index of Multiple Deprivation | 12 months
  Number of women attending cervical screening by level of deprivation (Scottish Index of Multiple Deprivation) (control vs intervention)
HPV vaccination status | 12 months
  Number of women attending cervical screening by HPV vaccination status (control vs intervention)

IPD SHARING:
Plan to Share IPD: No